CLINICAL TRIAL: NCT04736667
Title: Mitral Valve Screening Survey (MVSS)
Brief Title: Mitral Valve Screening Survey
Acronym: MVSS
Status: Recruiting | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MVSS
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Mitral Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects fail screening for TMVI: Subjects with symptomatic mitral valve disease who after referral for TMVI, are deemed not to be candidates for TMVI.

SUMMARY:
This study aims to examine the clinical profile/anatomical characteristics and natural history of patients who subsequently fail screening for transcatheter mitral valve intervention (TMVI).

DETAILED DESCRIPTION:
Numerous transcatheter mitral valve interventions have emerged as a treatment option for patients with mitral valve disease. Development of transcatheter mitral valve repair (TMVr) and transcatheter mitral valve replacement (TMVR) continues to progress with ongoing rigorous clinical trials of several experimental devices. However, despite being referred for TMVI, most patients do not pass stringent screening criteria for these investigational devices and are not offered TMVI.

In this prospective multicenter registry, baseline demographics, anatomical/imaging characteristics, and clinical outcomes of patients who fail screening for TMVI will be prospectively collected into a registry database.

ELIGIBILITY:
Inclusion Criteria:

* Subject failed screening for TMVI

Exclusion Criteria:

* Under 18 years of age
* Subject unable or unwilling to give informed consent
* Subject proceeded with TMVI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This multicenter prospective study will enroll consecutive subjects, who after referral for TMVI, are deemed not to be candidates for TMVI.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 1 year

SECONDARY OUTCOMES:
Reason for screen failure | Baseline
All-cause mortality | 30 days, 1 year, and annually up to 5 years
Hospitalizations | 30 days, 1 year, and annually up to 5 years
Mitral intervention | 30 days, 1 year, and annually up to 5 years

CONTACTS AND LOCATIONS:
Locations (16):
- United States (14):
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - Keck Hospital of USC, Los Angeles, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - HealthPark Medical Center, Fort Myers, Florida
  - Northwestern University, Chicago, Illinois
  - MercyOne Iowa Heart Center, West Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Ascension St. John's Hospital, Detroit, Michigan
  - NYU Langone Health - Long Island, Mineola, New York
  - The Ohio State University, Columbus, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Unity Health Toronto; St. Michael's Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Medranda GA, Rogers T, Modine T, Latib A, Jorde U, Bapat V, Sorajja P, Rowland M, Sutton JA, Baig S, Asch FM, Garcia-Garcia HM, Ben-Dor I, Satler LF, Waksman R. The Clinical Profile and Natural History of Patients Who Fail Screening for Transcatheter Mitral Valve Replacement: Rationale and Design of the Prospective Multicenter Mitral Valve Screening Survey (MVSS). Cardiovasc Revasc Med. 2023 Feb;47:72-75. doi: 10.1016/j.carrev.2022.09.003. Epub 2022 Sep 11. PMID 36266153
- [Derived] Waksman R, Medranda GA. Transcatheter Mitral Valve Replacement: Size Matters. JACC Cardiovasc Interv. 2021 Oct 25;14(20):2228-2230. doi: 10.1016/j.jcin.2021.08.040. Epub 2021 Sep 29. No abstract available. PMID 34600872